CLINICAL TRIAL: NCT03377439
Title: The Association Between Platelet Reactivity and Bleeding Risk in Adult ITP Patients: a Prospective Multicenter Double-blind Study
Brief Title: The Association Between Platelet Reactivity and Bleeding Risk in Adult ITP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Traditional Chinese Medicine Hospital Affiliated to Shandong University (Unknown); Jinan Central Hospital (Other); Qianfoshan Hospital (Other); Shandong Provincial Hospital (Other Government); Shandong University Second Hospital (Unknown)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Other Study IDs: Plt function and bleeding risk
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Immune Thrombocytopenia
Keywords: Platelet function; Bleeding risk; Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Platelet Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Participants with platelet counts <32×10^9/L.
  Interventions: Other: Platelet function tests
- Group B: Participants with platelet counts between 32×10^9/L and 132×10^9/L.
  Interventions: Other: Platelet function tests
- Group C: Participants with platelet counts >132×10^9/L.
  Interventions: Other: Platelet function tests

INTERVENTIONS:
Other: Platelet function tests — Platelet reactivity was measured by flow cytometry, filopodia detection and the platelet aggregation analyzer.

SUMMARY:
It seems reasonable to assume that patients who present significant bleeding symptoms may have different quality of platelets than those without bleeding. This question was addressed in a study that examined platelet function in adult ITP patients, which try to determine whether this correlated with bleeding risk. Previous reports have suggested that measuring platelet function may help define patients at highest risk of bleeding. In addition, Middelburg and colleagues corrected platelet function for quartile of platelet count, using <32×10^9/L as the lowest cohort and >132×10^9/L as the top quartile. They demonstrated that increased platelet reactivity (as measured by flow cytometry) was associated with decreased risk of bleeding but particularly for those patients with the lowest platelet counts. Further studies in a larger cohort are needed to confirm this correlation. Our study aimed at standardizing a prediction model to evaluate the bleeding risk of adult ITP patients with the use of platelet function tests.

DETAILED DESCRIPTION:
The investigators are undertaking a prospective multicenter double-blind study of 400 adult patients with immune thrombocytopenia from 6 medical centers in China. We adopted three different assays that examined platelet function and reactivity. 1) Flow cytometry: Citrate anticoagulated whole blood was diluted in PBS to result in 20×10^9/L platelets, and 20 μl was aliquoted into polystyrene test tubes. Ten microliters of anti-CD42b-PE was added and incubated at room temperature for 10 min. Agonists (TRAP-6 12.5 μMol/L, Collagen 20 μg/mL, ADP 2 μM, Epinephrin 20 μM, Arachidonic acid 0.275 mM, Ristocetin 1.5 mg/mL) or PBS were added (10 μl each) and incubated again for 10 min. Then mAb PAC-1-FITC or anti-CD62p-FITC (10 μl each) or the corresponding isotype-matched controls were added. After 15-min incubation in the dark, the reaction was stopped with 500 μl PBS. Samples were analyzed on a flow cytometer (FACScan, Becton-Dickinson) by measuring 10,000 events in the CD42b-positive fraction. 2) Filopodia quantification: Briefly, platelets in Tyrode's buffer were allowed to adhere to VWF (9×10^6 cells/coverslip) in the presence of botrocetin (1 μg/mL) and Integrilin (40 μg/mL) at 37°C. After 15 min, non-adherent platelets were removed by washing and adherent platelets were fixed with 4% PFA, stained with TRITC-phalloidin (2 μg/mL) and viewed by epifluorescence microscopy for filopodia count. 3) Platelet aggregation: Measured on an automated platelet aggregation analyzer.

Understanding bleeding risk and underlying determinants of bleeding is important in order to help recognize patients that will require pharmacologic therapy even at higher platelet counts. Previous studies have suggested that low platelet counts, increased patient age, use of concurrent medications, and male sex are associated with increased bleeding risk. The present investigation will answer whether platelet function predicts the severity of bleeding in adult ITP patients. Clinical information of recruited participants includes gender, age, platelet count and physical/laboratory examination. Blinding was set between investigators who evaluated bleeding risks and those who performed experiments.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated adult ITP patients of both genders between the ages of 18 and 80 years.
2. Participants of either acute or chronic phase; with or without thrombocytopenia; with or without bleeding manifestation.

Exclusion Criteria:

1. Received high-dose steroids or IVIG within 3 weeks prior to the test.
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months prior to the test.
3. Current HIV infection, hepatitis B virus or hepatitis C virus infections.
4. Severe medical condition (liver and kidney function impairment).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Untreated adult ITP patients of both genders between the ages of 18 and 80 years.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The severity of bleeding manifestations at onset was assessed using a previously described clinical scoring system with minor modifications. The total bleeding score was calculated by adding the scores for each item. | No more than three months after platelet function assessment.
  The bleeding score system: 1) Age: Age over 65 years (2'); Age over 75 years (5'). 2) Cutaneous bleeding: Localized petechial purpura (1'); Localized ecchymotic purpura (2'); Two locations of petechial purpura (2'); Generalized petechial purpura (3'); Generalized ecchymotic purpura (4'). 3) Mucosal bleeding: Unilateral epistaxis (2'); Bilateral epistaxis (3'); Hemorrhagic oral bullae and/or gingival bleeding (5'). 4) Gastrointestinal bleeding: Gastrointestinal hemorrhage without anemia (4'); Gastrointestinal hemorrhage with acute anemia and/or shock (15'). 5) Urinary bleeding: Macroscopic hematuria without anemia (4'); Macroscopic hematuria with acute anemia (10'). 6) Genitourinary tract bleeding: Major meno/metrorrhagia without anemia (4'); Major meno/metrorrhagia with acute anemia (10'). 7) Central nervous system bleeding: Central nervous system bleeding and/or life-threatening hemorrhage (15').

CONTACTS AND LOCATIONS:
Overall Officials: Jun Peng, MD, PhD, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khellaf M, Michel M, Schaeffer A, Bierling P, Godeau B. Assessment of a therapeutic strategy for adults with severe autoimmune thrombocytopenic purpura based on a bleeding score rather than platelet count. Haematologica. 2005 Jun;90(6):829-32. PMID 15951296
- [Background] Middelburg RA, Roest M, Ham J, Coccoris M, Zwaginga JJ, van der Meer PF. Flow cytometric assessment of agonist-induced P-selectin expression as a measure of platelet quality in stored platelet concentrates. Transfusion. 2013 Aug;53(8):1780-7. doi: 10.1111/trf.12001. Epub 2012 Dec 7. PMID 23216254
- [Background] Middelburg RA, Carbaat-Ham JC, Hesam H, Ragusi MA, Zwaginga JJ. Platelet function in adult ITP patients can be either increased or decreased, compared to healthy controls, and is associated with bleeding risk. Hematology. 2016 Oct;21(9):549-51. doi: 10.1080/10245332.2016.1180097. Epub 2016 May 9. PMID 27159138
- [Background] Panzer S, Hocker L, Koren D. Agonists-induced platelet activation varies considerably in healthy male individuals: studies by flow cytometry. Ann Hematol. 2006 Feb;85(2):121-5. doi: 10.1007/s00277-005-0029-5. Epub 2005 Nov 10. PMID 16283308
- [Background] Panzer S, Rieger M, Vormittag R, Eichelberger B, Dunkler D, Pabinger I. Platelet function to estimate the bleeding risk in autoimmune thrombocytopenia. Eur J Clin Invest. 2007 Oct;37(10):814-9. doi: 10.1111/j.1365-2362.2007.01855.x. Epub 2007 Aug 28. PMID 17727674
- [Background] Mangin P, Yuan Y, Goncalves I, Eckly A, Freund M, Cazenave JP, Gachet C, Jackson SP, Lanza F. Signaling role for phospholipase C gamma 2 in platelet glycoprotein Ib alpha calcium flux and cytoskeletal reorganization. Involvement of a pathway distinct from FcR gamma chain and Fc gamma RIIA. J Biol Chem. 2003 Aug 29;278(35):32880-91. doi: 10.1074/jbc.M302333200. Epub 2003 Jun 17. PMID 12813055
- [Background] Maurer E, Tang C, Schaff M, Bourdon C, Receveur N, Ravanat C, Eckly A, Hechler B, Gachet C, Lanza F, Mangin PH. Targeting platelet GPIbbeta reduces platelet adhesion, GPIb signaling and thrombin generation and prevents arterial thrombosis. Arterioscler Thromb Vasc Biol. 2013 Jun;33(6):1221-9. doi: 10.1161/ATVBAHA.112.301013. Epub 2013 Apr 4. PMID 23559635